CLINICAL TRIAL: NCT03383731
Title: A Single Center, Randomized and Controlled Clinical Study of Inverted Internal Limiting Membrane Insertion Combined With Air Tamponade in the Treatment of Macular Hole Retinal Detachment in High Myopia
Brief Title: A Study of a New Surgical Treatment of Macular Hole Retinal Detachment in High Myopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Fenghua Wang, Doctoral supervisor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shanghai1stWFH
Record Dates: First submitted 2017-12-06; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Macular Holes; Retinal Detachment; High Myopia
Keywords: Operation mode; Air tamponade; High myopia; Macular hole retinal detachment
MeSH Terms: conditions — Retinal Perforations; Retinal Detachment

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled study involving multiple visits within 12 months. The patients with macular hole retinal detachment caused by high myopia are randomly divided into 2 treatment groups.
  Group 1: standard 3-port 23 gauge pars plana vitrectomy + internal limiting membrane peeling + air-fluid exchange + silicone oil infusion Group 2: standard 3-port 23 gauge pars plana vitrectomy + internal limiting membrane peeling + inverted internal limiting membrane insertion + air-fluid exchange
Who Masked: Outcomes Assessor
Masking Description: In this study, the third party independent evaluation method is used to evaluate the results of the study. The analyzer is in the masking state, and the subjects and the surgeons are in the non-masking state..
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Group 1: The patients in Group 1 are treated by the surgical method of standard 3-port 23 gauge pars plana vitrectomy + internal limiting membrane peeling + air-fluid exchange + silicone oil infusion
  Interventions: Procedure: Group 1
- Group 2 (Experimental): Group 2: The patients in Group 2 are treated by the surgical method of standard 3-port 23 gauge pars plana vitrectomy + internal limiting membrane peeling + inverted internal limiting membrane insertion + air-fluid exchange
  Interventions: Procedure: Group 2

INTERVENTIONS:
Procedure: Group 1 — the surgical method of standard 3-port 23 gauge pars plana vitrectomy + internal limiting membrane peeling + air-fluid exchange + silicone oil infusion
  Arms: Group 1
Procedure: Group 2 — the surgical method of standard 3-port 23 gauge pars plana vitrectomy + internal limiting membrane peeling + inverted internal limiting membrane insertion + air-fluid exchange
  Arms: Group 2

SUMMARY:
This study evaluates the surgical outcomes of inverted internal limiting membrane insertion combined with air tamponade in the treatment of macular hole retinal detachment (MHRD) in high myopia, and also to compare the treatment efficacy and safety between different surgical approaches of MHRD

DETAILED DESCRIPTION:
This study uses a new surgical method (vitrectomy combined with inverted internal limiting membrane insertion and intraocular sterilized air tamponade) to assess its effectiveness and safety on the prognosis of macular hole retinal detachment secondary to high myopia, and also compares this new type of surgery with the current commonly used surgery (vitrectomy combined with internal limiting membrane peeling + silicone oil infusion).

ELIGIBILITY:
Inclusion Criteria:

1. Prior written informed consent should be obtained before any assessment is carried out;
2. Participants are more than 18 years of age, and less than 75 years of age, male or female Chinese patients;
3. Visual impairment is caused by macular hole associated with retinal detachment secondary to high myopia;
4. Axial length ≥ 26mm, or the refractive error ≥ -6.0D

Exclusion Criteria:

1. Failure to comply with research or follow-up procedures;
2. Diabetes with uncontrolled blood glucose (defined as fasting plasma glucose more than 7.0mmol/L or blood glucose more than 11.1mmol/ L 2 hours postprandial), and / or with diabetic retinopathy;
3. Poor control of blood pressure in hypertensive patients (defined as blood pressure >150/95mmHg, including antihypertensive medication);
4. With surgical contraindication due to other local or systemic conditions at screening or baseline;
5. With any active ocular or periocular infection or inflammation (e.g., blepharitis, conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) at screening or baseline;
6. With uncontrolled glaucoma at screening or baseline (IOP ≥ 30mmHg when receiving medical treatment or as judged by the researchers);
7. With the presence of iris neovascularization or neovascular glaucoma at screening or baseline;
8. With ocular diseases which may interfere the study results at screening or baseline , including severe vitreous hemorrhage, peripheral retinal hole, proliferative diabetic retinopathy, proliferative vitreoretinopathy ( ≥ Level C ), choroidal detachment;
9. With other causes which may result in macular hole associated-retinal detachment at screening or baseline,except high myopia;
10. Previously underwent scleral buckling surgery;
11. With current or planned medication known to have toxic effects on the lens, retina or optic nerve, including hydroxychloroquine, chloroquine, hydroxychloroquine, tamoxifen, phenothiazine and ethambutol;
12. With laboratory abnormalities, such as alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TB), gamma-glutamyl transferase (GGT), lactate dehydrogenase (LDH), exceeded the normal limit by more than 2 times, and serum creatinine or blood urea nitrogen exceeded 1.2 times the normal limit;
13. With abnormal coagulation function (defined as more than normal prothrombin time for 3 seconds or more, more than 1.5 of the international standard ratio (INR), activated partial thromboplastin time of 10 seconds or longer than the upper limit of normal time); 14) Patients who participated in any clinical study of medication within 3 months prior to screening (excluding vitamins and minerals)

Exit criteria:

1. Due to adverse events, especially severe adverse events, the researchers consider withdrawal of patients based on concerns of safety and ethics;
2. Drop out;
3. The patients voluntarily withdraw the informed consent;
4. Serious violation of the study protocol due to the subjects or investigators' reasons;
5. Other reasons that the researchers believe for quitting the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-04-07 (Actual); Primary Completion 2020-04-06 (Estimated); Study Completion 2020-04-06 (Estimated)

PRIMARY OUTCOMES:
Macular hole closure rate | 3 months after operation
  Fundus examination combined with optical coherence tomography (OCT) are performed 3 months after surgery.

SECONDARY OUTCOMES:
Best corrected visual acuity | 6 months after the operation
  Best corrected visual acuity are performed 6 months after the surgery.
Best corrected visual acuity | 12 months after the operation
  Best corrected visual acuity are performed 12 months after the surgery.
Reattachment rate of retinal detachment | 6 months after the operation
  Use fundus examination combined with B-scan ultrasound, optical coherence tomography (OCT) to observe the reattachment rate of retinal detachment within 12 months after the surgery.(The reattachment rate assessment is performed 12 months after the first surgery among the patients with air tamponade. The reattachment rate assessment is performed 12 months after the first surgery among the patients with silicone oil tamponade, and the silicone oil removal is performed 6 months after the previous surgery.)
Reattachment rate of retinal detachment | 12 months after the operation
  Use fundus examination combined with B-scan ultrasound, optical coherence tomography (OCT) to observe the reattachment rate of retinal detachment within 12 months after the surgery.(The reattachment rate assessment is performed 12 months after the first surgery among the patients with air tamponade. The reattachment rate assessment is performed 12 months after the first surgery among the patients with silicone oil tamponade, and the silicone oil removal is performed 6 months after the previous surgery.)
Postoperative complication rate of ocular adverse events | Within 12 months after operation
  Evaluate the ocular adverse events within 12 months after operation.
Postoperative complication rate of the non ocular adverse events | Within 12 months after operation
  Evaluate the non ocular adverse events within 12 months after operation.
Postoperative complication rate of severe adverse events | Within 12 months after operation
  Evaluate the severe adverse events within 12 months after operation.

OTHER OUTCOMES:
The number of people whose best corrected visual acuity (BCVA) result improves | 12 months after the operation
  The number of people whose BCVA result improves by more than 1 row, 2 rows and 3 rows comparing to the baseline at a time
The number of people whose BCVA result decreases | 12 months after the operation
  The number of people whose BCVA result decreases by 3 rows comparing to the baseline at a time
The difference of multifocal electroretinogram (ERG) results | 6 months after the operation
  The difference of multifocal ERG results between each group from 1 week to the 6th month after surgery
The difference of multifocal ERG results | 12 months after the operation
  The difference of multifocal ERG results between each group from 1 week to the 12th month after surgery
The change of microperimetry analysis results | 6 months after the operation
  The change of microperimetry analysis results from 1 week to the 6th month after surgery relative to baseline, and the difference between each group
The change of microperimetry analysis results | 12 months after the operation
  The change of microperimetry analysis results from 1 week to the 12th month after surgery relative to baseline, and the difference between each group
The change of the extent of foveal ellipsoid zone damage | 6 months after the operation
  The change of the extent of foveal ellipsoid zone damage from baseline to the 6th month after the surgery relative to baseline, and the difference between each group
The change of the external limiting membrane integrity of fovea | 6 months after the operation
  The change of the external limiting membrane integrity of fovea from baseline to the 6th month after the surgery relative to baseline, and the difference between each group
The change of the extent of foveal ellipsoid zone damage | 12 months after the operation
  The change of the extent of foveal ellipsoid zone damage from baseline to the 12th month after the surgery relative to baseline, and the difference between each group
The change of the external limiting membrane integrity of fovea | 12 months after the operation
  The change of the external limiting membrane integrity of fovea from baseline to the 12th month after the surgery relative to baseline, and the difference between each group
The number of retreatment and retreatment modalities | within 12 months after the operation
  λ Describe the number of retreatment and retreatment modalities for patients with different surgical procedures over a period of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fenghua Wang, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Statistical Analysis Plan that underlie results in a publication
Supporting Information: SAP
Time Frame: starting 6 months after publication
Access Criteria: Dr Fenghua Wang and Dr Ying Zheng will review requests and criteria.

REFERENCES:
- [Background] Feman SS, Hepler RS, Straatsma BR. Rhegmatogenous retinal detachment due to macular hole. Management with cryotherapy and a Y-shaped sling. Arch Ophthalmol. 1974 May;91(5):371-2. doi: 10.1001/archopht.1974.03900060383007. No abstract available. PMID 4595402
- [Background] Hong MC, Wu TT, Sheu SJ. Primary gas tamponade in the management of macular hole with retinal detachment in highly myopic eyes. J Chin Med Assoc. 2011 Mar;74(3):121-4. doi: 10.1016/j.jcma.2011.01.026. Epub 2011 Feb 25. PMID 21421206
- [Background] Miyake Y. A simplified method of treating retinal detachment with macular hole. Long-term follow-up. Arch Ophthalmol. 1986 Aug;104(8):1234-6. doi: 10.1001/archopht.1986.01050200140070. PMID 3741257
- [Background] Mete M, Parolini B, Maggio E, Pertile G. 1000 cSt silicone oil vs heavy silicone oil as intraocular tamponade in retinal detachment associated to myopic macular hole. Graefes Arch Clin Exp Ophthalmol. 2011 Jun;249(6):821-6. doi: 10.1007/s00417-010-1557-9. Epub 2010 Nov 16. PMID 21080197
- [Background] Soheilian M, Ghaseminejad AK, Yazdani S, Ahmadieh H, Azarmina M, Dehghan MH, Moradian S, Anisian A, Peyman GA. Surgical management of retinal detachment in highly myopic eyes with macular hole. Ophthalmic Surg Lasers Imaging. 2007 Jan-Feb;38(1):15-22. doi: 10.3928/15428877-20070101-02. PMID 17278531
- [Background] Li X, Wang W, Tang S, Zhao J. Gas injection versus vitrectomy with gas for treating retinal detachment owing to macular hole in high myopes. Ophthalmology. 2009 Jun;116(6):1182-87.e1. doi: 10.1016/j.ophtha.2009.01.003. Epub 2009 Apr 17. PMID 19375168
- [Background] Uemoto R, Yamamoto S, Tsukahara I, Takeuchi S. Efficacy of internal limiting membrane removal for retinal detachments resulting from a myopic macular hole. Retina. 2004 Aug;24(4):560-6. doi: 10.1097/00006982-200408000-00009. PMID 15300077
- [Background] Lim LS, Tsai A, Wong D, Wong E, Yeo I, Loh BK, Ang CL, Ong SG, Lee SY. Prognostic factor analysis of vitrectomy for retinal detachment associated with myopic macular holes. Ophthalmology. 2014 Jan;121(1):305-310. doi: 10.1016/j.ophtha.2013.08.033. Epub 2013 Oct 16. PMID 24139155
- [Background] Shin MK, Park KH, Park SW, Byon IS, Lee JE. Perfluoro-n-octane-assisted single-layered inverted internal limiting membrane flap technique for macular hole surgery. Retina. 2014 Sep;34(9):1905-10. doi: 10.1097/IAE.0000000000000339. No abstract available. PMID 25154029
- [Background] Michalewska Z, Michalewski J, Dulczewska-Cichecka K, Adelman RA, Nawrocki J. TEMPORAL INVERTED INTERNAL LIMITING MEMBRANE FLAP TECHNIQUE VERSUS CLASSIC INVERTED INTERNAL LIMITING MEMBRANE FLAP TECHNIQUE: A Comparative Study. Retina. 2015 Sep;35(9):1844-50. doi: 10.1097/IAE.0000000000000555. PMID 25946691
- [Background] Kuriyama S, Hayashi H, Jingami Y, Kuramoto N, Akita J, Matsumoto M. Efficacy of inverted internal limiting membrane flap technique for the treatment of macular hole in high myopia. Am J Ophthalmol. 2013 Jul;156(1):125-131.e1. doi: 10.1016/j.ajo.2013.02.014. Epub 2013 Apr 24. PMID 23622567
- [Background] Hasegawa Y, Hata Y, Mochizuki Y, Arita R, Kawahara S, Kita T, Noda Y, Ishibashi T. Equivalent tamponade by room air as compared with SF(6) after macular hole surgery. Graefes Arch Clin Exp Ophthalmol. 2009 Nov;247(11):1455-9. doi: 10.1007/s00417-009-1120-8. Epub 2009 Jun 21. PMID 19544065
- [Background] He F, Dong F, Yu W, Dai R. Recovery of photoreceptor layer on spectral-domain optical coherence tomography after vitreous surgery combined with air tamponade in chronic idiopathic macular hole. Ophthalmic Surg Lasers Imaging Retina. 2015 Jan;46(1):44-8. doi: 10.3928/23258160-20150101-07. PMID 25559508
- [Background] Mateo-Montoya A, de Smet MD. Air as tamponade for retinal detachments. Eur J Ophthalmol. 2014 Mar-Apr;24(2):242-6. doi: 10.5301/ejo.5000373. Epub 2013 Sep 23. PMID 24170524
- [Derived] Zheng Y, Kang M, Wang H, Liu H, Sun T, Sun X, Wang F. Inverted internal limiting membrane insertion combined with air tamponade in the treatment of macular hole retinal detachment in high myopia: study protocol for a randomized controlled clinical trial. Trials. 2018 Aug 30;19(1):469. doi: 10.1186/s13063-018-2833-y. PMID 30165894

DOCUMENTS (2):
  • Informed Consent Form (2017-04-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT03383731/ICF_000.pdf
  • Study Protocol (2017-04-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT03383731/Prot_001.pdf